CLINICAL TRIAL: NCT03069027
Title: Efficacy of External Nasal Nerve Block on Postoperative Agitation Following Nasal Surgeries Under General Anesthesia. Randomized, Controlled Trial
Brief Title: Efficacy of External Nasal Nerve Block in Prevention of Postoperative Agitation Following Nasal Surgeries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al Jedaani Hospital (Other)
Responsible Party: Principal Investigator, Dr. Mohamed Ibrahim, Assistant Professor of Anesthesiology- Zagazig University - Consultant of anesthesia, Al Jedaani Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 3-2-17
Record Dates: First submitted 2017-02-19; First posted 2017-03-03 (Actual); Last update posted 2017-12-27 (Actual); Status verified 2017-12

CONDITIONS: Agitation States as Acute Reaction to Gross Stress
Keywords: Nasal surgery; external nasal nerve block; postoperative agitation
MeSH Terms: interventions — Lidocaine; Epinephrine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group I(control) (Placebo Comparator): patients allocated for external nasal nerve block with saline adrenaline 1/200,000 (placebo)
  Interventions: Procedure: External nasal nerve block; Drug: saline adrenaline
- Group II(block) (Active Comparator): 'External nasal nerve block by Xylocaine, adrenaline'
  Interventions: Procedure: External nasal nerve block; Drug: Xylocaine, adrenaline

INTERVENTIONS:
Procedure: External nasal nerve block — Three single (midline injection) and 4 paired (bilateral injection) sites to block the external nasal sensation.
Drug: saline adrenaline
  Arms: Group I(control)
Drug: Xylocaine, adrenaline
  Arms: Group II(block)

SUMMARY:
Emergence agitation following general anaesthesia may lead to serious complications like self-extubation or removal of catheters, which can lead to hypoxia, aspiration pneumonia, bleeding or reoperation. Nose surgery is associated with a higher incidence of emergence agitation. The investigators planned to evaluate the efficacy of external nasal nerve block in prevention of postoperative agitation following external nasal surgeries under general anesthesia(GA).

ELIGIBILITY:
Inclusion Criteria:

* 110 adult patients of ASA physical status I and II,
* Age 20-60 years,
* Scheduled for elective external nasal surgeries in which nasal packing on each side was used postoperatively for 24 hours.

Exclusion Criteria:

1. History of uncontrolled hypertension,
2. Ischemic or valvular heart disease,
3. Use of MAO inhibitors or adrenergic blocking drugs,
4. Cognitive impairment,
5. Patients taking antipsychotics,
6. Renal insufficiency or liver dysfunction

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2016-08-15 (Actual); Primary Completion 2017-04-15 (Actual); Study Completion 2017-07-01 (Actual)

PRIMARY OUTCOMES:
postoperative agitation | Emergence is defined as the time interval from discontinuation of anesthesia to 5 min after extubation.
  Assessment done using Richmond agitation- sedation scale (RASS)
Quality of recovery | 24 hours postoperative
  Quality of recovery

SECONDARY OUTCOMES:
dose of fentanyl | intraoperative period in minutes
  Fentanyl boluses were given in response to changes in hemodynamics (more than 15% increases in MAP and HR than the baseline values taken after induction by 5 minutes)
morphine dose in PACU | one hour in PACU
  equivalent morphine dose in PACU (calculated using opioid:morphine equivalents of 100 µg i.v. fentanyl to 10 mg i.v. morphine; 75- 100 mg IV pethidine to 10 mg i.v. morphine
Nausea and vomiting in PACU | one hour in PACU
  Four-point nausea and vomiting scale (0=no nausea; 1=mild nausea; 2=severe nausea requiring antiemetics; and 3=retching, vomiting, or both) was also evaluated
Extubation time | Up to 15 after discontinuation of anesthesia
Surgical time | duration of surgery in minutes up to 3 hours
  intraoperative
first verbal response time | up to 15 minutes
  period from discontinuation of anesthesia 'time zero' to 1st verbal response in minutes
complication of nasal block | From injection to 24 hours postoperative
  including local anesthetic systemic toxicity, vascular injury, intravascular injection of local anesthetic, and local hematoma.

CONTACTS AND LOCATIONS:
Locations (1):
- Al Jedaani group of hospitals, Jeddah, Meccah, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided